CLINICAL TRIAL: NCT04667039
Title: International, Multicenter, Randomized, Double-blind, Comparative Clinical Study of the Efficacy, Safety, Pharmacokinetics, and Immunogenicity of GNR-067 and Lucentis® in Patients With Neovascular (Wet) Age-related Macular Degeneration
Brief Title: Efficacy, Safety, pharmacokinetiсs, Immunogenicity of GNR-067 and Lucentis®
Acronym: NAP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: AO GENERIUM (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RBS-AMD-III
Record Dates: First submitted 2020-11-30; First posted 2020-12-14 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Age Related Macular Degeneration (ARMD)
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

STUDY DESIGN:
Intervention Model Description: Interventional
Who Masked: Investigator
Masking Description: Throughout the study, until the end of the comparative treatment study period, neither the investigators nor the patients knew which drug was being administered
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GNR-067 (Experimental): Ranibizumab
  Interventions: Biological: Lucentis®
- Lucentis® (Active Comparator): Ranibizumab
  Interventions: Biological: GNR-067

INTERVENTIONS:
Biological: GNR-067 — GNR-067 will be used intravitreally once every 4 weeks in 0.5 mg doses (the injection volume is 0.05 mL)
  Other Names: Ranibizumab
  Arms: Lucentis®
Biological: Lucentis® — Lucentis® will be used intravitreally once every 4 weeks in 0.5 mg doses (the injection volume is 0.05 mL)
  Other Names: Ranibizumab
  Arms: GNR-067

SUMMARY:
This is a randomized, double-blind, comparative, parallel group study of the efficacy, safety pharmacokinetics, and immunogenicity of GNR-067 and Lucentis® in patients with neovascular (wet) age-related macular degeneration.

DETAILED DESCRIPTION:
Age-related macular degeneration (ARMD) is a chronic progressive disease that is the main cause of visual disability in elderly patients (aged over 60 years) in industrialized countries. Due to increased human longevity, it is expected for the number of patients with this disease to grow worldwide up to 288 million people by 2040. The highest risk of vision loss is posed by neovascular (exudative or wet ARMD) macular degeneration observed in 10-20% of cases. The pathological changes of ARMD are based on the increased production of the vascular endothelial growth factor (VEGF) which affects proprioceptors located on the surface of endothelial cells and causes an anomalous permeability of vessels and stimulates neovascularization GNR-067 (JSC "GENERIUM", the Russian Federation) is a humanized recombinant monoclonal antibody selectively binding to the human vascular endothelial growth factor [VEGF-A] and is a biosimilar of of the original product Lucentis® ("Novartis Pharma AG", Switzerland).

This III phase study is aimed to compare the effectiveness, safety, pharmacokinetics and immunogenicity of GNR-067 (JSC "GENERIUM", the Russian Federation) and Lucentis® ("Novartis Pharma AG", Switzerland) in order to register of the drug GNR-067 (JSC "GENERIUM", the Russian Federation), a solution for intraocular injection administration, in the Russian Federation.

The study included patients (n = 408) aged 50 years and older with neovascular (wet) age-related macular degeneration, types 1 and 2 (occult and classical) choroidal neovascularization (CNV) with the following activity signs: accumulation of intraretinal and/or subretinal (under the neurosensory retina or pigment epithelium) fluid, extravasal dye exit from the newly formed vessels, and the presence of a subfoveal and/or juxtafoveal membrane and the presence of CNV foci of more than 50% of the total lesion area. With block randomization, the patients were divided into two groups in a 2:1 ratio (investigational/reference product): 272 patients to the group of the investigational product GNR-067 and 136 patients to the group of the reference product Lucentis®. The duration of the study for each patient will be approximately 52 ± 4 weeks, including a screening period (3 weeks), treatment period and a follow-up period (4 weeks). In this study GNR-067 and Lucentis® will be used intravitreally once every 4 weeks (thirteen injections in total) in 0.5 mg doses (the injection volume is 0.05 mL).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 50 years and older;
2. The signed informed consent obtained from the patient, or, in cases of severe visual impairment in the patient, with the participation of an impartial witness, prior to any study-related procedures.

   Ophthalmic inclusion criteria (must be present in one eye, which will be considered the examined eye)
3. The previously diagnosed neovascular (wet) age-related macular degeneration confirmed at the Screening Visit:

   untreated, except for food supplement, vitamins, mineral additives (one examined eye in one patient); Types 1 and 2 (occult and classical) choroidal neovascularization (CNV) with the following activity signs: accumulation of intraretinal and/or subretinal (under the neurosensory retina or pigment epithelium) fluid, extravasal dye exit from the newly formed vessels, and the presence of a subfoveal and/or juxtafoveal membrane and the presence of CNV foci of more than 50% of the total lesion area;
4. The best-corrected visual acuity within a range from 34 to 83 letters (20/200 to 20/25) measured using the ETDRS chart Early Treatment Diabetic Retinopathy Study Research Group protocol (chart at a distance of 4 m) before pupil dilation;
5. The willingness and ability of the patient to perform all planned study visits and procedures (according to the Investigator);
6. IOP ≤21 mmHg (actual);
7. An ECG within normal values or clinically insignificant findings.

Exclusion Criteria:

1. Medical history of CNV treatment with intravitreal injections of VEGF inhibitors (ranibizumab, bevacizumab, aflibercept, or pegaptanib, etc.), or any other investigational poducts into the examined eye;
2. Medical history of subretinal laser photocoagulation or other surgical interventions for ARMD in any eye;
3. Preexisting and current lesions, diseases, or interventions in the eyes.:

   In the examined eye:

   Keratoplasty or corneal dystrophy Capsulotomy performed 4 weeks prior to screening Aphakia, vitrectomy Presence of a macular hole at any stage Past rhegmatogenous retinal detachment Any other past intraocular surgical interventions in the examined eye (including cataract extraction in the examined eye) within 3 months prior to the Screening Visit

   In any eye:

   Choroidal neovascularization in any eye due to reasons not related to ARMD (for example, multifocal choroiditis, ocular histoplasmosis syndrome, injury, etc.) Past idiopathic or autoimmune uveitis in any eye Scleromalacia Diagnosed diabetic retinopathy

   Current conditions and diseases identified at the screening stage:

   High degree myopia (over 8 diopters) in any eye; Presence of progressive glaucoma (intraocular pressure ≥21 mmHg against performed antihypertensive glaucoma therapy) or optic neuropathy that affect or endanger the central field of view in the examined eye at the screening stage; Subretinal hemorrhage and/or hemorrhage in the retinal tissue occupying ≥50% of the total affected area in the examined eye; Presence of a rupture (solution of continuity) of the retinal pigment epithelium (RPE) also extending to the macula in any eye; A scar or subretinal fibrosis in the macular area occupying more than 50% of the total affected area in any eye; Presence of vitreomacular traction or epiretinal membrane significantly affecting central vision; Other than ARMD progressive retinal diseases in the examined or fellow eye that may complicate the assessment of visual acuity; The total size of the lesion is more than 12 disc areas (DA: 30.5 mm2 including areas occupied by blood, neovascularization, or fibrosis), based on a FAG performed at screening; Confirmed or assumed (within 28 days prior to the Screening Visit) intraocular, extraocular, and periocular inflammation or infection in any eye.
4. Any intravitreal injections of corticosteroids (e.g., triamcinolone acetonide) for ≥30 days in a row in the examined eye 90 days prior to the Screening Visit and/or injection of an intravitreal corticosteroid implant with a gradual release of the medicinal product into the examined eye within 180 days prior to the Screening Visit;
5. Known allergic reactions and/or hypersensitivity to Lucentis® (ranibizumab) or any ingredients of GNR-067;
6. Known allergic reactions and/or hypersensitivity to fluorescein sodium (for injections);
7. Uncontrolled arterial hypertension (BP ≥180/90 mmHg);
8. Diseases of the immune and endocrine system, not controlled by drug therapy (including decompensated diabetes mellitus and thyroid diseases);
9. Medical history or current (active cancer)of oncological diseases with the exception of cured basal cell carcinoma;
10. Vaccination (any vaccine) within 30 days prior to the Screening Visit and/or the need for vaccination during the study period;
11. Systemic treatment with corticosteroids (more than 10 mg of prednisolone equivalent) within 6 months prior to the Screening Visit;
12. Use of systemic medicinal products known to be toxic for the eye lens, retina, or optic nerve during the study.
13. Medical history of a clinically significant pathology identified during the screening period including, but not limited to:

    Unstable angina pectoris, myocardial infarction, arrhythmia requiring drug therapy, Class III or IV congestive heart failure according to the New York Heart Association classification within one year before the Screening Visit; Brain injury, stroke, or transient ischemic attack within one year prior to the Screening Visit; Severe renal failure (estimated glomerular filtration rate according to the CKD-EPI formula <40 mL/min/1.73 m2); Severe hepatic impairment (serum alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) activity of 2.5 or more times higher than the laboratory upper limit of normal (ULN), and/or the level of total bilirubin of 1.5 or more times higher than the laboratory ULN);

    Variation of peripheral blood parameters:

    Leukocytes: <3.8 × 109/L Platelets: <100 × 109 cells/L Hemoglobin: ≥10.0 g/dL
14. Pregnancy and breastfeeding;
15. Patients who received blood or blood component transfusions within 10 days prior to the Screening Visit;
16. History (within three years prior to the Screening Visit) of tuberculosis, alcoholism, narcotic, drug dependence and/or substance abuse, or presence of the above at the Screening stage;
17. Acute hepatitis or liver cirrhosis of any etiology; antibodies to hepatitis C or HBsAg at the Screening Visit; acquired immune deficiency syndrome or infection with human immunodeficiency virus (HIV) confirmed by test results;
18. Participation of the patient in any clinical studies and/or use of experimental medicinal products within 3 months prior to the Screening Visit.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2022-03-20 (Actual); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients (%) with an increase in the best-corrected visual acuity (BCVA) score on the ETDRS chart (measured using logMAR/Snellen chart) of 15 or more letters at Week 8 versus baseline in the compared groups. | At 8 Week after comparative treatment beginning (GNR-067 vs. Lucentis®).
  Global evaluation of treatment effectiveness (the best-corrected visual acuity (BCVA) score on the ETDRS chart (measured using logMAR/Snellen chart)) of 15 or more letters are a validated tool and has been used to evaluate the clinical response to ranibizumab in patients with with neovascular (wet) age-related macular degeneration.

SECONDARY OUTCOMES:
The proportion of patients (%) with an increase in the best-corrected visual acuity (BCVA) score on the ETDRS chart (measured using logMAR/Snellen chart) of 15 or more letters at Week 24, Week 52 versus baseline in the compared groups. | At Week 24, Week 52 after comparative treatment start (GNR-067 vs. Lucentis®) and compared to baseline.
  The best-corrected visual acuity (BCVA) score on the ETDRS chart (measured using logMAR/Snellen chart)) of 15 or more letters are a validated tool and has been used to evaluate the clinical response to ranibizumab in patients with with neovascular (wet) age-related macular degeneration.
The proportion of patients (%) with a decrease in the best-corrected visual acuity (BCVA) score on the ETDRS chart (measured using logMAR/Snellen chart) of 15 or fewer letters at Week 8, Week 24, and Week 52 versus baseline in the compared groups. | At Week 8, Week 24, Week 52 weeks after comparative treatment start (GNR-067 vs. Lucentis®) and compared to baseline.
  The best-corrected visual acuity (BCVA) score on the ETDRS chart (measured using logMAR/Snellen chart) of 15 or fewer letters are a validated tool and has been used to evaluate the clinical response to ranibizumab in patients with with neovascular (wet) age-related macular degeneration.
The decrease of the central retinal thickness (CRT) measured with optical coherence tomography in the spectral range at Week 8, Week 24, Week 52 versus baseline in the compared groups. | At Week 8, Week 24, Week 52 versus baseline in the compared groups.
  The decrease of the central retinal thickness (CRT) in patient with neovascular (wet) age-related macular are standard of the optical coherence tomography (OCT).
The proportion of patients (%) with the presence (incomplete recovery) of intraretinal fluid and subretinal fluid at Week 8, Week 24, Week 52 versus baseline in the compared groups. | At Week 8, Week 24, Week 52 versus baseline in the compared groups
  The presence (incomplete recovery) of intraretinal fluid and subretinal fluid in patient with neovascular (wet) age-related macular are standard for fluorescent angiography.
The assessment of changes in visual acuity and quality of life of patients by the questionnaire method using the NEI VFQ-25 medical ophthalmological questionnaire at Week 24 Week 52 versus baseline in the compared groups. | At Week 24 Week 52 versus baseline in the compared groups.
  NEI VFQ-25 medical ophthalmological questionnaire is standard of the assessment changes in visual acuity and quality of life of patients with neovascular (wet) age-related macular.
Immunogenicity | The frequency of formation of ADAs to ranibizumab at Day 1, Day 8, Week 8, Week 24, Week 36, and Week 52 of treatment with the investigational or reference product with the characterization of antibodies.
  The frequency of antidrug antibodies formation.

CONTACTS AND LOCATIONS:
Overall Officials: Oksana Markova, MD, Study Chair — AO GENERIUM
Locations (9):
- Russia (9):
  - Regional budgetary healthcare institution "Ivanovo Regional Clinical Hospital", Ivanovo, Ivanovo Oblast
  - State Budgetary Healthcare Facility of the St. Petersburg Region "First St. Petersburg State Medical University named after academician I.P. Pavlova "of the Ministry of Health of the Russian Federation, Saint Petersburg, Leningradskaya Oblast'
  - Federal State Budgetary Educational Institution of Higher Education "Moscow State University of Medicine and Dentistry named after A.I. Evdokimov "of the Ministry of Health of the Russian Federation, Moscow, Moscow Oblast
  - Federal State Autonomous Institution "Interbranch Scientific and Technical Complex" Eye Microsurgery "named after academician S.N. Fedorov "of the Ministry of Health of the Russian Federation, Moscow, Moscow Oblast
  - State Budgetary Healthcare Institution of the Novosibirsk Region "State Novosibirsk Regional Clinical Hospital", Novosibirsk, Novosibirsk Oblast
  - State Budgetary Healthcare Institution of the Omsk region "Clinical ophthalmological hospital named after V.P. Vykhodtseva", Omsk, Omsk Oblast
  - State Autonomous Healthcare Institution "Republican Clinical Ophthalmological Hospital of the Ministry of Health of the Republic of Tatarstan" Kazan, Kazan', Tatarstan Republic
  - Limited Liability Company "Kuzlyar", Kazan', Tatarstan Republic
  - Federal State Budgetary Educational Institution of Higher Education "Samara State Medical University" of the Ministry of Health of the Russian Federation, Kazan', Tatarstan Republic

IPD SHARING:
Plan to Share IPD: No
NAP